CLINICAL TRIAL: NCT00704340
Title: DuraSeal Sealant Post Market Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DRS-05-002
Record Dates: First submitted 2008-06-23; First posted 2008-06-24 (Estimated); Results first posted 2010-07-28 (Estimated); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Elective Cranial Procedures With Dural Incision
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): DuraSeal Dural Sealant System - FDA Approved Device:
  The DuraSeal™ Dural Sealant System is a polyethylene glycol (PEG) hydrogel that has been FDA approved as a dural sealant to achieve watertight dural closure in cranial and spinal surgery after primary repair with suturing is complete. It was developed as a means of providing a dural seal by covering small holes around the suture with an absorbable hydrogel.
  Interventions: Device: DuraSeal Dural Sealant System
- 2 (Active Comparator): Standard of Care (control):
  Standard procedure to obtain intraoperative watertight dural closure. These methods could have included additional sutures, adhesive glue, absorbable gelatin sponge, dural substitute, soft tissue patch, or another method typically used by the investigator.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: DuraSeal Dural Sealant System — The DuraSeal™ Dural Sealant System is a polyethylene glycol (PEG) hydrogel that has been FDA approved as a dural sealant to achieve watertight dural closure in cranial and spinal surgery after primary repair with suturing is complete. It was developed as a means of providing a dural seal by covering small holes around the suture with an absorbable hydrogel. DuraSeal should only be used with autologous duraplasty material.
  Arms: 1
Other: Standard of Care — Standard procedure to obtain intraoperative watertight dural closure. These methods could have included additional sutures, adhesive glue, absorbable gelatin sponge, dural substitute, soft tissue patch, or another method typically used by the investigator.
  Other Names: Standard procedure to obtain intraoperative watertight dural closure
  Arms: 2

SUMMARY:
DuraSeal Dural Sealant has been approved as a dural sealant by the FDA for use in cranial and spinal procedures. This study was completed to further evaluate the safety of the DuraSeal Sealant in a post-approval setting as compared to control (defined as methods typically employed by surgeons to seal the dura).

ELIGIBILITY:
Inclusion Criteria:

* Patient is between 18 and 75 years of age
* Patient is scheduled for an elective cranial procedure that entails a dural incision
* Evidence of intraoperative non-watertight closure

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2005-09; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Confluent Surgical, Waltham, Massachusetts, United States

REFERENCES:
- [Derived] Osbun JW, Ellenbogen RG, Chesnut RM, Chin LS, Connolly PJ, Cosgrove GR, Delashaw JB Jr, Golfinos JG, Greenlee JD, Haines SJ, Jallo J, Muizelaar JP, Nanda A, Shaffrey M, Shah MV, Tew JM Jr, van Loveren HR, Weinand ME, White JA, Wilberger JE. A multicenter, single-blind, prospective randomized trial to evaluate the safety of a polyethylene glycol hydrogel (Duraseal Dural Sealant System) as a dural sealant in cranial surgery. World Neurosurg. 2012 Nov;78(5):498-504. doi: 10.1016/j.wneu.2011.12.011. Epub 2011 Dec 10. PMID 22381303

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject was enrolled on September 12, 2005, last subject visit was May 20, 2009.
Pre-assignment Details: Randomized study, no washout or run-in period.
Groups:
- DuraSeal: DuraSeal Dural Sealant System - FDA Approved Device
- Control: Standard of Care (control)
Period: Overall Study
Arm/Group | DuraSeal | Control
Started | 120 | 117
Completed | 118 | 115
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | DuraSeal | Control | Total
Number analyzed (Participants) | 120 | 117 | 237
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 108 | 102 | 210
  >=65 years | 12 | 15 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.6 (14.1) | 48.2 (13.5) | 48.9 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 74 | 152
  Male | 42 | 43 | 85
Region of Enrollment [Number; unit: participants]
  United States | 120 | 117 | 237

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Surgical Wound Complications, Central Nervous System Events, and Neurosurgical Complications Related to Unplanned Intervention or Return to the Operating Room.
Description: Surgical Wound Complications;
  * Superficial incisional surgical site infection (SSI)
  * Deep incisional SSI
  * Organ/Space SSI
  * Late incisional infection: superficial incisional infection that occurs more than 31 but less than 38 days after surgery
  * Poor wound healing
  Central Nervous System Events;
  * Cerebrospinal Fluid (CSF) leak
  * Hydrocephalus
  * Bacterial meningitis
  * Aseptic meningitis
  In addition, any complication related to the neurosurgical procedure that required unplanned intervention (i.e., minimally invasive procedures) or return to the operating room was counted.
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percent of subjects
Arm/Group | DuraSeal | Control
Number analyzed (Participants) | 120 | 117
percent of subjects | 5.8 [2.4 to 11.6] | 7.7 [3.6 to 14.1]
Statistical Analysis 1: Comparison: DuraSeal vs Control; The sample size was selected to provide sufficient precision for 95% confidence intervals for the incidence of neurosurgical complications in each arm. The sample size was selected so that the half-width of the normal approximation-based intervals would be no more than 0.05 percentage points. This requires a sample size of 114 evaluable patients in each arm. To allow for loss to follow-up, the sample size was increased to 125 randomized patients in each treatment arm, or a total of 250 patients; Test type: Superiority or Other; p = .613, t-test, 2 sided

2. Secondary Outcome: Percentage of Subjects With Post-operative Surgical Site Infections
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percent of subjects
Arm/Group | DuraSeal | Control
Number analyzed (Participants) | 120 | 117
percent of subjects | 1.7 [.2 to 5.9] | 2.6 [.5 to 7.3]
Statistical Analysis 1: Comparison: DuraSeal vs Control; Test type: Superiority or Other; p = .681, t-test, 2 sided

3. Secondary Outcome: Percentage of Subjects With a Cerebrospinal Fluid (CSF) Leak
Description: As determined from clinical diagnosis by one of the following methods:
  * CSF leak or pseudomeningocele related surgical intervention (i.e., breaking skin) within 30 days post-operation
  * CSF leak confirmation by diagnostic testing within 30 days post-operation
  * CSF leak confirmation by clinical evaluation including physical examination of the surgical site within 30 days post-operation
Time Frame: 30 days
Measure: Number (95% Confidence Interval); unit: percent of subjects
Arm/Group | DuraSeal | Control
Number analyzed (Participants) | 120 | 117
percent of subjects | 0.8 [0 to 4.6] | 1.7 [.2 to 6.0]
Statistical Analysis 1: Comparison: DuraSeal vs Control; Test type: Superiority or Other; p = .619, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | DuraSeal | Control
Serious Adverse Events (participants affected / at risk) | 15/120 | 19/117
Other Adverse Events (participants affected / at risk) | 0/120 | 0/117
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DuraSeal (N=120) | Control (N=117)
Acute Gait Dysfunction/Readmission (Nervous system disorders) | 1 (1) | 0 (0)
evacuation of epidural hematoma (Nervous system disorders) | 1 (1) | 0 (0)
pulmonary embolus (Cardiac disorders) | 0 (0) | 2 (2)
C. Difficile (Infections and infestations) | 0 (0) | 1 (1)
Transient Ischemic Attack (T.I.A.) (Cardiac disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 3 (3)
Deep Incisional SSI (Infections and infestations) | 2 (2) | 0 (0)
Superficial Incisional SSI (Infections and infestations) | 0 (0) | 3 (3)
Headache and intractable nausea/vomiting (Nervous system disorders) | 0 (0) | 1 (2)
Headache (Nervous system disorders) | 3 (3) | 0 (0)
Cerebrovascular Accident (C.V.A.)- also known as stroke (Cardiac disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pancreatitis (General disorders) | 0 (0) | 1 (1)
Cerebral hemmorhage (Nervous system disorders) | 3 (3) | 1 (1)
Malignant Metastatic melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Blood clot (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aseptic meningitis (Infections and infestations) | 0 (0) | 1 (1)
Central diabetes insipidus (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
CSF leak (Nervous system disorders) | 1 (1) | 1 (1)
Late incisional SSI (Infections and infestations) | 1 (1) | 0 (0)
headache/double-vision (Nervous system disorders) | 0 (0) | 1 (1)
left hemiplegia (Nervous system disorders) | 1 (1) | 0 (0)
nausea/vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
cerebral vasospasm (Nervous system disorders) | 0 (0) | 1 (1)
Bacteremia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
cerebral edema (Nervous system disorders) | 1 (1) | 0 (0)
brain tumor (Nervous system disorders) | 1 (1) | 0 (0)
severe neurological deficit post-op (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less